CLINICAL TRIAL: NCT05574738
Title: An Exploratory Biomarker Analysis in Blood, Urine, Stools, Hair Follicles and Saliva of Patients With Malignant Disease
Brief Title: A Study to Explore Biomarkers in Samples of Blood, Urine, Stools, Hair Follicles and Saliva From Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: Eileen Soulis (Other)
Responsible Party: Sponsor-Investigator, Eileen Soulis, Project Manager, Cancer Research UK, Glasgow
Organization: Cancer Research UK, Glasgow (Other)
Other Study IDs: MI84_ECMC
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational

SUMMARY:
The goal of this observational study is to learn about biomarkers in patients with certain types of malignant solid tumours (cancer). The main intentions are to analyse changes in biomarkers before and after treatment, determine their relationship to how a tumour responds to treatment, and potentially identify new biomarkers or genetic markers to diagnose or predict disease.

Participants will be asked to provide additional samples of blood, urine, stools, hair follicles or saliva (depending on which type of cancer they have).

DETAILED DESCRIPTION:
This is a study in patients with confirmed malignant disease (solid tumour) due to start anti-cancer therapy/radiotherapy or attending for clinical assessment. Patients will be asked to give additional blood, hair, urine or saliva samples for research compared to standard treatment in this proposal. Blood (25 mL) will be taken, once, prior to starting therapy (or at routine assessment). Further samples of 25 mL of venous blood will be taken at each subsequent visit for chemotherapy in patients who undergo chemotherapy treatment, and at fixed timepoints for those undergoing treatment with non-chemotherapy regimens.

These timepoints will coincide with routine hospital visits for disease assessment purposes for these patients and no additional visits will be required. Similarly, a 20 mL sample of urine will be collected at the above timepoints from patients with urological cancers. A 2 mL sample of saliva will be collected at the above timepoints from patients with head and neck cancers. Where possible 25 mL of venous blood will also be collected at each subsequent follow-up visit after completion of chemotherapy (other systemic therapies, or radiation therapy) until there is documented disease progression. Patient treatment, supportive care and disease assessment will be unaffected by participation in this study. Collected samples will be analysed for biomarkers (proteins or DNA from tumour cells sometimes detected in a sample of blood or urine) at the Translational Pharmacology Lab, University of Glasgow. These biomarker results will be compared with patient outcome (objective response and overall survival) with the aim of developing biomarkers that might help us to better select the type of chemotherapy regimen given to individual patients. For patients with breast cancer who will be treated in the neo-adjuvant setting, they will be asked to provide 3 stool samples (prior to treatment, halfway through treatment and at the end of treatment) to study changes to gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed malignant disease (solid tumour) or a diagnosis of malignant disease made using recognised clinical criteria.
2. Patients who are attending for clinical assessments at presentation; during a routine hospital visit for anti-cancer therapy, radiotherapy, surgery, or for whom no immediate specific therapy is planned; or at a follow-up hospital visit.
3. Written informed consent.
4. Age ≥18 years.
5. Able to comply with study protocol.

Exclusion Criteria:

(1) Any evidence of any medical or psychiatric disorders that would, in the opinion of the investigator, be a contra indication to venesection, urine, stool or saliva collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant disease identified at clinical assessment at outpatient clinics or wards, either at presentation or when they are about to undergo anti-cancer therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-06-28 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Collect blood and/or, where appropriate, urine, hair, stool or saliva samples from patients with solid tumours | Before, during and immediately after therapeutic interventions.
  to analyse changes in the blood proteome, nucleic acids, faecal microbiome and in novel blood or urine or faecal or hair follicle or saliva biomarkers, during anti-cancer treatment in patients with malignant disease.
Collect blood and/or, where appropriate, urine, hair, stool or saliva samples from patients with solid tumours | Before, during and immediately after therapeutic interventions.
  to determine if baseline values of these markers, and/or changes during anti-cancer treatment, correlate with tumour response and / or treatment-related adverse events.
Collect blood and/or, where appropriate, urine, hair, stool or saliva samples from patients with solid tumours | Before therapeutic interventions.
  Novel prognostic, predictive and pharmacodynamic markers in blood (or urine or stool or hair follicles or saliva) of patients with early or advanced disease baseline: pre-intervention
Collect blood and/or, where appropriate, urine, hair, stool or saliva samples from patients with solid tumours | During therapeutic interventions
  Novel prognostic, predictive and pharmacodynamic markers in blood (or urine or stool or hair follicles or saliva) of patients with early or advanced disease baseline: during therapeutic interventions
Collect blood and/or, where appropriate, urine, hair, stool or saliva samples from patients with solid tumours | Immediately after therapeutic interventions
  Novel prognostic, predictive and pharmacodynamic markers in blood (or urine or stool or hair follicles or saliva) of patients with early or advanced disease baseline: immediately after therapeutic interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Evans, Prof, Principal Investigator — Cancer Research UK, Glasgow
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided